CLINICAL TRIAL: NCT05687526
Title: A Phase 1, Open-label, Multi-center, Multiple-dose Study to Evaluate the Pharmacokinetics of Telitacicept in Subjects With Childhood-onset Systemic Lupus Erythematosus
Brief Title: A Study of Telitacicept in Subjects With Childhood-onset Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18C018
Record Dates: First submitted 2023-01-08; First posted 2023-01-18 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: systemic lupus erythematosus; pediatrics; PK
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — telitacicept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telitacicept (Experimental): The dosing of Telitacicept frequency was based on body weight and age.
  Interventions: Biological: Telitacicept

INTERVENTIONS:
Biological: Telitacicept — 12-17 years old: Telitacicept 2.5 mg/kg (with a maximum dose of 160 mg) subcutaneously once a week plus SOC for 12 weeks.
  5-11years old: Telitacicept 3.0-3.5 mg/kg (with a maximum dose of 160 mg) subcutaneously once a week plus SOC for 12 weeks.
  Other Names: RC18

SUMMARY:
This is a multi-center, open-label, phase 1 study.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the pharmacokinetics (PK) of multiple doses of Telitacicept in subjects with childhood-onset systemic lupus erythematosus (cSLE) on a background of standard of care therapy and explore the safety and efficacy of Telitacicept in patients with cSLE.

ELIGIBILITY:
Main Inclusion Criteria:

1. Fulfills SLICC 2012 or 2019 EULAR/ACR classification criteria for SLE.
2. 5-17 years of age when signing the informed consent.
3. Suject and/or legal guardian or parent provided written informed consent.
4. SELENA SLEDAI score ≥ 8 at screening.
5. Serum autoantibodies (ANA and/or anti ds-DNA) tested positive at screening.
6. Have been on a stable standard of care for SLE for at least 30 days prior to randomization.
7. Female patients are required to be non-pregnant, non-lactating or sterile.

Main Exclusion Criteria:

1. Have received Telitacicept at any time.
2. Have received any of the following therapies within 6 months of baseline: B-cell targeted treatment, e.g., belimumab, rituximab, abatacept, other investigational biologicals.
3. Have received any of the following therapies within 90 days of baseline: anti-TNF or anti-IL-6 therapy, interleukin-1 receptor antagonist, intravenous immunoglobulin (IVIG), plasmapheresis.
4. Have received any of the following therapies within 30 days of baseline: Intravenous cyclophosphamide, non-biological investigational agents (within 30 days of baseline or 5 half-lives, whichever is longer), newly added immunosuppressive/immunomodulatory agent, anti-malarial, NSAID, high-dose prednisone or equivalent (> 1.5 mg/kg/day) or any intramuscular or intravenous steroid.
5. Have received live vaccine within 30 days of baseline.
6. Participated in an interventional clinical trial within 6 months of screening.
7. Active CNS lupus requiring treatment within 60 days of baseline, including seizure, psychosis, organic brain syndrome, cerebrovascular accident, cerebritis or CNS vasculitis.
8. Currently on kidney replacement therapy (hemodialysis, peritoneal dialysis) or in need of such therapy within 90 days of baseline.
9. eGFR<30 mL/min/1.73m2.
10. Acute severe nephritis.
11. History of vital organ transplant (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/marrow transplant.
12. Significant unstable or uncontrolled acute or chronic diseases (cardiovascular, lung, hematology, gastrointestinal, liver, renal, neurologic, malignancy or infectious disease) that could be explained by causes other than SLE.

13 Have planned surgery, laboratory abnormalities, other diseases or conditions that, in the opinion of the investigator, makes the subject unsuitable for the study.

14. History of malignant neoplasm in the past 5 years. 15. Primary immune deficiency. 16. Acute or chronic infections requiring treatment. 17. HIV or HCV positive. 18. Tuberculosis. 19.HBsAg/HbcAb positive. 20.HBcAb positive. 21.History of COVID-19 within 4 weeks prior to screening. 22.History of hospitalization due to severe Covid-19 within 12 months prior to screening.

23.History of allergy to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies.

24.History of drug or alcohol abuse or dependence within 364 days prior to baseline.

25.Investigators believe that there are other factors that are not suitable for participating in the experiment.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Cmax of Telitacicept | up to 42 days following the last dose of Telitacicept
  Cmax is defined as peak plasma concentration of Telitacicept
tmax of Telitacicept | up to 42 days following the last dose of Telitacicept
  tmax is defined as time to reach Cmax of Telitacicept
Ctrough of Telitacicept | up to 42 days following the last dose of Telitacicept
  Ctrough is defined as observed plasma concentration of Telitacicept just prior to the beginning of a dosing interval
Cav of Telitacicept | up to 42 days following the last dose of Telitacicept
  Average concentration of Telitacicept
AUC0-t of Telitacicept | up to 42 days following the last dose of Telitacicept
  AUC0-t is defined as area under the curve from time zero to last quantifiable concentration of Telitacicept
t1/2z of Telitacicept | up to 42 days following the last dose of Telitacicept
  t1/2z is defined as terminal elimination half-life of Telitacicept
λz of Telitacicept | up to 42 days following the last dose of Telitacicept
  λz is defined as terminal elimination rate constant

SECONDARY OUTCOMES:
SLE Responder Index 4 (SRI 4) | Week 4, Week 8, Week 12
  SRI 4 is defined as a. SELENA-SLEDAI score reduced from baseline by at least 4 points; b. no new BILAG A or no more than 1 BILAG B compared to baseline; c. physician's global assessment (PGA) increased from baseline by less than 0.3 points.
Proportion of subjects with SELENA-SLEDAI score reduced from baseline by at least 4 points. | Week 4, Week 8, Week 12
  The SELENA-SLEDAI is a tool for measuring the activity of systemic lupus. The total score ranges from 0-105, with a higher score representing a more significant degree of disease activity.
Change from baseline in PGA. | Week 4, Week 8, Week 12
  The PGA is a visual analog scale scored from 0 to 3. A score of 1 corresponds to mild lupus disease activity. A score of 2 correlates with moderate disease activity and a score of 3 with severe disease activity.
Change From Baseline in IgG | Week 4, Week 8, Week 12
  Immunoglobulins (IgG, IgA and IgM) are proteins produced by plasma cells.
Change From Baseline in IgA | Week 4, Week 8, Week 12
  Immunoglobulins (IgG, IgA and IgM) are proteins produced by plasma cells.
Change From Baseline in IgM | Week 4, Week 8, Week 12
  Immunoglobulins (IgG, IgA and IgM) are proteins produced by plasma cells.
Change From Baseline in C3 | Week 4, Week 8, Week 12
  Complement (C3/C4) are proteins that are part of the immune system.
Change From Baseline in C4 | Week 4, Week 8, Week 12
  Complement (C3/C4) are proteins that are part of the immune system.
Incidence of AEs | up to Week 12
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hongmei Song, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (12):
- China (12):
  - Children's Hospital of Capital Institute of Pediatrics, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Henan Children's Hospital, Zhengzhou, Henan
  - Hunan Children's Hospital, Changsha, Hunan
  - Nanjing Children's Hospital, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Xi'an Children's Hospital, Xi'an, Shaanxi
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Chengdu Women's & Children's Central Hospital, Chengdu, Sichuan
  - Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided